CLINICAL TRIAL: NCT04577950
Title: A Prospective Phase 2 Study Comparing Three Injection Sites to Detect Sentinel Lymph Nodes in Endometrial Cancer: Comparison of Lymphatic Drainages and Location of the Sentinel Lymph Nodes Depending on the Injection Site of the Tracer
Brief Title: A Prospective Study Comparing Three Injection Sites to Detect Sentinel Lymph Nodes in Endometrial Cancer
Acronym: SENNAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, prof. Patrice Mathevet, Head of the gynecologic department, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SENNAN
Record Dates: First submitted 2020-09-12; First posted 2020-10-08 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Endometrial Cancer
Keywords: Sentinel node; Endometrial carcinoma; Lymphatic drainage
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective phase 2 study comparing three injection sites to detect sentinel lymph nodes in endometrial cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm with procedure: identification of lymphatic drainage of the uterus following 3 sites injections (Experimental): A radiocolloid (Nanocoll® marked with Technetium 99), a fluorochrome (ICG) and a blue dye (Bleu Patenté®) will be injected in submucosal tissue to see the differences in lymphatic drainage between three different injection sites. Indeed, ICG will be injected under the endometrium, whereas Nanocoll® will be injected in the cervix and Bleu Patenté® in the uterine isthmus, at the transition between the cervix and the uterine corpus.
  Interventions: Procedure: Lymphatic drainage of endometrial cancer

INTERVENTIONS:
Procedure: Lymphatic drainage of endometrial cancer — Nanocoll® is injected a day before surgery in the cervix at four points. A lymphoscintigraphy is performed 2 or 3 hours afterward. At the beginning of the surgery, the operative field already in place and before the beginning of laparoscopic, 2ml (10mg) of ICG, distributed in four points around the tumor, is injected under the endometrium intra-myometrial under endoscopic control. As ICG spreads slower than blue dye, ICG is always injected first. Then, Bleu Patenté® is injected at two sites in the uterine isthmus, opposite of the uterine arteries. The risk of false negative results, because a tracer migrated too quickly, is reduced when the injection takes place when patients are already anesthetized.

SUMMARY:
Uterine cancer is the most common gynecologic malignancy in developed countries. Adenocarcinoma of the endometrium is the most common histologic type of uterine cancer. Endometrial cancer is the fifth most frequent cancer in women in Switzerland. The incidence rose up to 5.9% in 2015. This tumor affects mainly older women, at 63 years on average. The majority of women are diagnosed at an early stage. Seventy-five to 90% of the patients are alerted by abnormal uterine bleeding very quickly, which allows a quick management of care and a high survival rate.

Besides age, one of the main risk factor of developing an endometrial carcinoma is obesity. In fact, obese women have higher risk to have an endometrial cancer, but also at a younger age than the average and finally they have an increased risk of death due to this particular cancer. Although this cancer is linked to the co-morbidities that go with obesity like diabetes or hypertension.

The treatment of endometrial cancer in most women is surgery involving a total hysterectomy and a bilateral salpingo-oophorectomy with or without a lymph node dissection. For patients with early stage endometrial cancer, there is a disagreement regarding lymph nodes dissection, because randomized controlled trials and a meta-analysis have shown no clear evidence on overall or recurrence-free survival and a higher incidence on early and late complications in relation with pelvic lymph node dissection. A systematic lymph node dissection consists of removing all the nodes within a nodal drainage basin. This dissection proves to be very difficult in obese patient and includes a risk to damage blood vessels or nerves. Moreover, lymph node dissection is associated with a higher morbidity, longer operating time, more frequent blood loss and finally symptomatic lymphedema and seroma.

That is why, sentinel lymph node biopsy (SLNB) seems to be a good alternative to lymph node dissection. The tumor's spread is assessed in lymph nodes with a reduced morbidity. In fact, lymphadenectomy and its dangerous complications, like lymphedema, could be avoided in the vast majority of cases. Indeed, a histological analysis of these sentinel lymph-nodes (SLNs) leads to ultrastadification: cancers are graded depending on the presence and the size of metastasis in lymph nodes. Adjuvant treatments, such as radiotherapy or chemotherapy, can be suggested following these data and a better management of endometrial cancer is possible.

DETAILED DESCRIPTION:
Worldwide, in 2012, 527'600 women were diagnosed with uterine cancer. It is the most common gynecologic malignancy in developed countries. In developing countries, it is the second most common, just behind cervical cancer. Adenocarcinoma of the endometrium is the most common histologic site and type of uterine cancer. Endometrial cancer is the fifth most frequent cancer in women in Switzerland. The incidence rose up to 5.9% in 2015. This tumor affects mainly older women, at 63 years on average. The majority of women are diagnosed at an early stage: confined to primary site for 67%, spread to regional organs and lymph nodes for 21% and with distant metastasis for 8%. Seventy-five to 90% of the patients are alerted by abnormal uterine bleeding very quickly, which allows a quick management of care and a high survival rate.

Besides age, one of the main risk factor of developing an endometrial carcinoma is obesity. In fact, obese women have higher risk to have an endometrial cancer, but also at a younger age than the average and finally they have an increased risk of death due to this particular cancer. Although the investigators are not sure of the reasons, it may be linked to the co-morbidities that go with obesity like diabetes or hypertension.

The treatment of endometrial cancer in most women is surgery involving a total hysterectomy and a bilateral salpingo-oophorectomy with or without a lymph node dissection. For patients with early stage endometrial cancer, there is a disagreement among cancer centers regarding lymph nodes dissection, because randomized controlled trials and a meta-analysis have shown no clear evidence on overall or recurrence-free survival and a higher incidence on early and late complications in relation with pelvic lymph node dissection. A systematic lymph node dissection consists of removing all the nodes within a nodal drainage basin irrespective of size. The problem with that technique is that dissection proves to be very difficult in obese patient and includes a risk to damage blood vessels or nerves.Moreover, lymph node dissection is associated with a higher morbidity, longer operating time, more frequent blood loss and finally symptomatic lymphedema and seroma. Indeed, the risk of leg lymphedema due to a node dissection is often under-reported, with rates going from 5% to 38%.

That is why, sentinel lymph node biopsy (SLNB) seems to many authors to be a good alternative to lymph node dissection. The tumor's spread is assessed in lymph nodes with a reduced morbidity. In fact, lymphadenectomy and its dangerous complications, like lymphedema, could be avoided in the vast majority of cases. In cutaneous melanoma or in breast's cancer, this technique is already widely used throughout the world. A sentinel node is the first node involved in the movement of the tumor from the primary cancer to the lymph nodes. When tumor cells spread to lymphatic network, they arrive in the first place in that sentinel node. If it contains no metastasis, then nodes, on the lymph path below, will not be affected either.

Not only SLNB in endometrial cancer is associated with a reduction in morbidity compared to lymph node dissection, but with it, a personalized treatment can be developed. Indeed, a histological analysis of these sentinel lymph-nodes (SLNs) leads to ultrastadification: cancers are graded depending on the presence and the size of metastasis in lymph nodes. Adjuvant treatments, such as radiotherapy or chemotherapy, can be suggested following these data and a better management of endometrial cancer is possible. Now, when lymph-node status is still unknown, indication for adjuvant therapies are based on pathological features of surgical specimens of the tumor, exposing some patients to either overtreatment or undertreatment.

In fact, five-year disease free survival in stage I patients with positive SLNs is 54%, whereas survival with negative SLNs is up to 90%.Therefore, SLN is one of the most important prognostic factors in endometrial cancer.

Primary objective of SENNAN study: The study seeks primarily to compare the location of uterine SLNs depending on the injection sites of the tracers: whether in endometrium, in uterine isthmus or in the cervix.

Secondary objectives are:

1. A comparison of the sensitivity of the tracers to detect SLNs
2. A description of the incidence of adverse events
3. An evaluation of additional time required to identify SLNs with or without lymph node dissection.
4. A description of morbidity directly induced by the search of SLNs
5. A calculation of negative predictive value of the different markers and their associations
6. A correlation between the anatomical locations of the SLNs and ultrastadification of SLNs.
7. An evaluation of the data of the lymphatic drainage, depending on tumor location in the uterus.
8. An evaluation of the data of the lymphatic drainage, depending on histological grade of the tumor.
9. An analysis of cases wherein change in the treatment have been made related to results of detection of SLNs.

Procedure:

The patients will have the day before the surgery an identification of the sentinel nodes with radiocolloid (Nanocoll®). The marker at a radioactivity of 80 MBq will be injected in four points in the cervix, 0.2 ml of 20 millibecquerel each. A CTscintigraphy will be performed three or four hours after the injection. The day of the surgery, the patients will undergo a general anaesthesia and then under general anaesthesia, the first step of the surgery will be to do the injection of the other two markers :

* ICG® will be injected through hysteroscopic guidance apart of the tumoral lesions at 4 points of injections. The volume of injected ICG will be 0.5 ml at each injection at the concentration of 5 mg/ml. A total of 2 ml (10mg) of ICG will be used.
* Patent blue® will be diluted with 2 ml of physiologic serum. Then it will be injected through the cervix along the uterus isthmus at the 3 o'clock and 9 o'clock level. 2 ml will be injected on each side.

Then the patients will have a laparoscopic surgical approach with identification of the sentinel nodes in the pelvic and lower abdomen areas. After identification of all the sentinel nodes : blue and / or radioactive and / or fluorescent nodes, the patients will have a total hysterectomy with bilateral oophorectomy and salpingectomy. The surgical technique for this procedure is the same as the one usually performed for this kind of lesions.

The major benefit of looking for SLNs in endometrial cancer is that lymphadenectomy can be avoided for patients who have already comorbidities. Indeed, endometrial cancer is found in aged women and obese women are also more affected. Lymphadenectomy is a heavy procedure with a risk of lymphedema. That is why the technique of SLNs offers a good alternative with lesser surgical risks.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Early endometrial cancers (of International Federation of Gynecology and Obstetrics stage IA-IB), whatever histological grade and type
* Primary surgical treatment with hysterectomy
* No metastasis, no other cancers, no recurrency of cancers
* No signs of lymph nodes metastasis on the preoperative workup (MRI +/- positron emission computed tomography)
* No contraindication to laparoscopic procedures.
* Women of > 18 years

Exclusion Criteria:

* Known severe allergies (antecedents of Quincke oedema, anaphylactic shock,…) and a history of allergy to iodides
* Contraindications to the injected products because of known hypersensitivity or allergy to ICG of blue dye
* Antecedent of pelvic lymph nodes surgery
* Previous lymphadenectomy or surgery that could change the uterine lymphatic drainage (conisation or myomectomy)
* Other diagnosed cancer during treatment or care
* Stage II and above (tumor invading cervix stroma) including those after a neo-adjuvant treatment
* Suspicion of lymph nodes metastasis at preoperative workup
* Medical or uterine conservative treatment
* Patient, who does not understand, speak or write in French
* Drugs that can interfere with ICG : anti convulsants - bisulphite compounds - haloperidol - heroin - pethidine [meperidine] - methamizole - methadone - morphine - nitrofurantoin - opium alkaloids - phenobarbitone- phenylbutazone - cyclopropane - probenecid - rifamycin - sodium bisulphite (mostly combined with heparin)
* Radioactive iodine uptake performed less than one week following the use of ICG.
* Hypersensitivity to Nanocoll, to any of the excipients (Stannous chloride, dihydrate Glucose, anhydrous Poloxamer 238 Sodium phosphate, dibasic, anhydrous Sodium phytate, anhydrous) or to any of the components of the labelled radiopharmaceutical.
* A history of hypersensitivity to products containing human albumin
* Hypersensitivity to dyes made of triphenylmethane
* Lymphostasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Lymphatic route of endometrial cancer dissemination | 1 month
  Comparing the per-operative anatomical locations of uterine SLNs depending on the 3 different injection sites of the tracers: whether in endometrium, in uterine isthmus or in the cervix.

SECONDARY OUTCOMES:
Sensibility/sensitivity of the tracers | 1 month
  A comparison of the sensibility/sensitivity of the tracers to detect SLNs
Adverse events | 1 month
  A description of the incidence of adverse events
Additional time required to identify SLNs | 1 month
  An evaluation of additional time required to identify SLNs with or without lymph node dissection.
Morbidity directly induced by the search of SLNs | 1 month
  A description of morbidity grades (following the NCI CTCAE classification) directly induced by the search of SLNs
Negative predictive value of the different markers | 1 month
  A calculation of negative predictive value of the different markers and their associations
Correlation between the per-operative anatomical locations of the SLNs and ultrastadification of SLNs. | 1 month
  A correlation between the per-operative anatomical locations of the SLNs and the results of ultrastadification of these SLNs.
Comparison between the results of lymphatic drainage and location of the tumor. | 1 month
  An evaluation of the anatomical location of the SLNs depending on uterine location of the tumor.
  The anatomical locations would be divided in 3 different sites: pelvic, para-aortic and parametrial.
  The location of the tumor would be divided in 3 sites: uterine horns, uterine fundus, uterine walls.
Comparison between the results of lymphatic drainage and grade of the tumor. | 1 month
  An evaluation of the anatomical location of the SLNs depending on grade of the tumor.
  The anatomical locations would be divided in 3 different sites: pelvic, para-aortic and parametrial.
  The location of the tumor would be divided in 3 grades: 1, 2 and 3
Cases with change in treatment in relation with SLNs detection and histology. | 1 month
  Description of cases wherein change in the treatment have been made related to results of different anatomical locations and pathological (including ultrastadification) results of SLNs.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Mathevet, MD - PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUV department of gynecology, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All data will be accessed under request to the PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years
Access Criteria: Request to PI